CLINICAL TRIAL: NCT01478932
Title: Diaphragmatic Breathing Retraining in Heart Failure Patients: Health-Behavior Related Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left University
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0541-11-EP; 5P20NR011404-03 (NIH)
Record Dates: First submitted 2011-11-04; First posted 2011-11-23 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Dyspnea
Keywords: dyspnea; diaphragmatic breathing; Heart failure
MeSH Terms: conditions — Dyspnea; Heart Failure | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic Breathing Retraining (Experimental): In-person and written instructions will be given as to how to carry out the breathing retraining at home. Four telephone calls will be made from a member of the research team during the 8-week intervention at weeks 1, 2, 4, and 6. During the phone calls, progress and difficulties related to the breathing intervention will be discussed. A daily log to track performance of the intervention will be kept.
  Interventions: Behavioral: diaphragmatic breathing retraining
- Health Promotion (Placebo Comparator): In-person instructions will be given about what the intervention includes. Four telephone calls will be made from a member of the research team during the 8-week intervention at weeks 1, 2, 4, and 6. During the phone calls, health promotion topics will be discussed (lipid profile, healthy eating to improve lipid profile, importance of regular doctor visits, cancer screening, and so forth).
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: diaphragmatic breathing retraining — In-person and written instructions will be given as to how to carry out the breathing retraining at home. Four telephone calls will be made from a member of the research team during the 8-week intervention at weeks 1, 2, 4, and 6. During the phone calls, progress and difficulties related to the breathing intervention will be discussed. A daily log to track performance of the intervention will be kept.
  Arms: Diaphragmatic Breathing Retraining
Behavioral: Health Promotion — n-person instructions will be given about what the intervention includes. Four telephone calls will be made from a member of the research team during the 8-week intervention at weeks 1, 2, 4, and 6. During the phone calls, health promotion topics will be discussed (lipid profile, healthy eating to improve lipid profile, importance of regular doctor visits, cancer screening, and so forth).
  Arms: Health Promotion

SUMMARY:
The purpose of this study is to provide information on how the practicing of diaphragmatic breathing retraining (DBR) for 8-week at home may improve the health outcomes and encourage heart failure patients to engage in health-promoting activities by successfully controlling their shortness of breath (dyspnea).

DETAILED DESCRIPTION:
In heart failure (HF) patients, dyspnea is a key contributor to and the strongest predictor for hospital readmission. In addition, dyspnea and fatigue are the primary reasons for decreased physical activity (PA) which, in turn, leads to activity avoidance, subsequent muscle de-conditioning, and further increases of dyspnea even at lower levels of activity. Depression, because of its moderate relationship with dyspnea, can further diminish PA and increase disability in activities of daily living (ADLs). Strategies to minimize or mitigate dyspnea and to boost motivation are imperative for improving adherence to PA, and, in turn, improving fatigue, muscle strength, PA itself, functional status, disability in ADLs including basic ADLs and instrumental ADLs (IADLs), depression, and quality of life (QOL) in HF patients. The overall purpose of this pilot/feasibility study is to evaluate an 8-week, home-based DBR intervention, in HF patients who are experiencing dyspnea at rest or with daily activities. Using an experimental randomized controlled design, 50 participants over 19 years of age, with diagnosed with chronic HF, who experience dyspnea at rest or with activity and experience dyspnea that limits their activities, who have a telephone, and who reside in a rural area, will be recruited at the University of Nebraska Medical Center HF clinic and at the Veterans Affairs Nebraska-Western Iowa Hospital, Cardiology-Congestive Heart Failure clinic. Both groups will receive the usual care from a HF specialist. The experimental group will receive information on a Diaphragmatic Breathing Retraining (DBR) intervention whereas the health promotion (attention control) group will receive general health information. To boost adherence to the intervention and to prevent attrition from the study, both groups will receive telephone calls from a research nurse for a total of 4 sessions (weeks 1, 2, 4 and 6). During follow-ups via phone calls for the attention control group, the research personnel will discuss health promotion topics (e.g., lipids profile, health eating, cancer screening, and annual check-ups (e.g., flu shot, eye and/or dental exams) with their primary health care provider. Data collection using standardized measures, will take place at baseline, post-intervention, and 3-month follow-up after completion of the 8-week intervention. The primary outcomes are: dyspnea and fatigue. The secondary outcomes are: muscle strength, PA, functional status, depression, disability in ADLs, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. adults age 19 or older
2. diagnosed with chronic heart failure
3. experiencing shortness of breath at rest or with activities
4. experiencing shortness of breath that limits their activity
5. cognitively intact indicated by being able to describe what participation in the study will involve
6. have a telephone; AND
7. reside in a rural area either large rural (10,000-49,000 residents), small rural (2500- 9999 residents), or isolated (< 2499 residents) area

Exclusion Criteria:

1. myocardial infarction or coronary bypass surgery within the last three months
2. active chest pain
3. uncontrolled arrhythmias (atrial fibrillation or ventricular tachycardia)
4. on the transplant list or having a ventricular assist device
5. orthopedic or neurological conditions that would impact muscle strength or interfere with the 6- minute walk test (6-MWT) (amputation, severe arthritis, Parkinson's, stroke, or severe neuropathy)
6. history of severe chronic obstructive pulmonary disease (COPD); AND
7. history of sleep breathing disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-11-09 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Dyspnea | day 1, after 8-week intervention, after 5 months
  Dyspnea rating scale of 0 to 4 (0 = none to 4 = extraordinary)
Fatigue | day 1, after 8-week intervention, after 5 months
  Patient Reported Outcomes Measurement Information System (PROMIS-57) Profile fatigue scale of 0 to 5 (0 = not at all to 5 = very much)

SECONDARY OUTCOMES:
Muscle Strength | day 1, after 8-week intervention, after 5 months
  Muscle strength will be measured by a Nicholas hand held dynamometer with the participant seated in a chair with feet on the floor. Measuring hip extensors will be done in a standing position. Muscle strength will be measured in kilograms (kg) of the maximum force exerted by the participant. The participants will be asked to "push as hard as you can against the dynamometer."
Physical activity | day 1, after 8-week intervention, after 5 months
  Measured by placement of ActiHeart (Trade Mark) accelerometer monitor on participant in the morning and removal in the evening (times of placement and removal recorded in diary).
Functional Status (6 minute walk test) | day 1, after 8-week intervention, after 5 months
  A 6-minute walking test is conducted on a 20 meter (22 yard) long course in an enclosed corridor. A chair will be placed at each end of the course to mark the turnaround point. Participants will be asked to walk the course at their own pace, covering as much distance as comfortable. Participants may slow down or stop and rest during the walk but will be asked to resume the exercise as soon as able.
Functional Status (Timed Get Up & Go) | day 1, after 8-week intervention, after 5 months
  The participant will be asked to walk a distance of 3 meters along a line that will be timed at seconds from getting up from the chair, walking, and returning to sitting down in a chair.
Depression Inventory | day 1, after 8-week intervention, after 5 months
  Participants complete Beck Depression Inventory questionnaire consisting of 21 groups of statements concerning depression and respond from 0 (do not agree) to 3 (strongly agree).
Disability in Activities of Daily Life (ADL) | day 1, after 8-week intervention, after 5 months
  Participants complete Disabilities in ADL questionnaire of 7 activities of daily life and respond from 0 (need another person to do that on my behalf) to 3 (do it without assistance).
Quality of Life questionnaire (self-care, usual activities, pain/discomfort, & Anxiety/Depression) | day 1, after 8-week intervention, after 5 months
  Participants complete EuroQol Group EuroQual_5DL questionnaire of 5 daily activities/conditions and respond from no problem, some problem, unable to perform/extreme condition.

CONTACTS AND LOCATIONS:
Overall Officials: Yaewon Seo, PhD, Principal Investigator — University of Nebraska; Bernice Yates, PhD, Study Director — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States